CLINICAL TRIAL: NCT02528097
Title: A Randomized Comparison of Two Albumin Administration Schedules for Spontaneous Bacterial Peritonitis
Brief Title: A Comparison of Two Albumin Administration Schedules for Spontaneous Bacterial Peritonitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-00743
Record Dates: First submitted 2014-04-04; First posted 2015-08-19 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator Standard Care (Placebo Comparator): albumin administered day 1 (1.5g/kg) and day 3 (1.0g/kg)
  Interventions: Drug: Standard Care
- Experimental (Experimental): Albumin administered per standard care on day 1 (1.5g/kg). Second dose administered on day 2 only to those individuals with renal insufficiency and risk for renal failure (Cr > 1.0 or BUN or Cr > baseline). If albumin not administered at 48 hours, BUN and Cr will be monitored daily for 72 hours and will be administered if Cr > 1.0 or BUN or Cr are above baseline.
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Standard Care — Standard Care: 25% salt poor albumin administered day 1 (1.5g/kg) and day 3 (1.0g/kg)
  Arms: Active Comparator Standard Care
Drug: Experimental — 25% salt poor albumin administered per standard care on day 1 (1.5g/kg). Second dose administered on day 2 or later only to those individuals with renal insufficiency and risk for renal failure (Cr > 1.0 or BUN or Cr > baseline)
  Arms: Experimental

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a common and frequently fatal complication of end-stage liver disease with a mortality of up to 10% primarily due to the development of kidney failure. Current standard practice is to treat this infection with broad spectrum antibiotics and salt-poor albumin administration on day one and three of treatment. In this study the investigators test the hypothesis that the administration of a second dose of albumin at 48 hours only to patients with renal insufficiency is as effective at preventing kidney failure as administering the second dose to all patients at 72 hours. In addition, a kidney function determined approach to albumin dosing may lead to substantial cost and resource saving from decreased albumin use without compromising treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75
* Evidence of end stage liver disease / cirrhosis
* Documented SBP (ANC > 250 or positive ascites culture
* Ability to provide informed consent
* Serum Creatinine > 1.0 mg/dL and/or Total Bilirubin > 4.0 mg/dL

Exclusion Criteria:

* Nonportal hypertensive ascites (i.e. malignancy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Comparator Standard Care | Experimental
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator Standard Care | Experimental | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Renal Failure
Description: Primary outcome is the presence of renal failure at any point from the start of the study (time 0) through 72 hours
Time Frame: At any point from time 0 through day 3
Population: Outcome data was not collected due to logistical challenges of completing the study.
Arm/Group | Active Comparator Standard Care | Experimental
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: All Cause Mortality
Time Frame: At any point from time 0 through day 3
Population: Outcome data was not collected due to logistical challenges of completing the study.
Arm/Group | Active Comparator Standard Care | Experimental
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Administration of Albumin
Description: The amount of albumin administered to each study participant over the course of the study (time 0 through 72 hours)
Time Frame: Throughout Study (72 hours)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Active Comparator Standard Care | Experimental
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Due to the extremely small sample size, and the fact that the PI left the institution, no data was analyzed for this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes